CLINICAL TRIAL: NCT03052205
Title: A Phase 1b Study of Intratumoral IMO-2125 in Patients With Refractory Solid Tumors (ILLUMINATE-101)
Brief Title: A Study of Intratumoral IMO-2125 in Patients With Refractory Solid Tumors
Acronym: ILLUMINATE-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2125-RST-101
Record Dates: First submitted 2017-02-06; First posted 2017-02-14 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Refractory Solid Tumors; Melanoma
Keywords: ILLUMINATE-101; melanoma
MeSH Terms: conditions — Melanoma | interventions — tilsotolimod

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMO-2125 at escalating dose levels (Experimental): IMO-2125 at escalating dose levels by intratumoral injection
  Interventions: Drug: IMO-2125

INTERVENTIONS:
Drug: IMO-2125 — IMO-2125 will be administered by intratumoral injection on Days 1, 8, and 15 of Cycle 1 and on Day 1 of each subsequent cycle.

SUMMARY:
This is a Phase 1b study that incorporates dose expansion cohorts to further evaluate promising clinical or biological activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed diagnosis of cancer not amenable to curative therapy.
2. Patients who have a diagnosis for which a PD-(L)-1 inhibitor has been approved must have previously received treatment with one of these therapies.

   a. Melanoma Dose Expansion: Patients must have histologically confirmed metastatic melanoma (ocular melanoma not included) which has progressed on or after treatment with a PD-(L)1 inhibitor.
3. a) Dose Evaluation Portion: Patients should have at least one lesion accessible for intratumoral injection and biopsy.

   b) Melanoma Expansion Cohort: Patients must have at least one target lesion by Response Evaluation Criteria for Solid Tumors (RECIST v1.1), with at least one lesion accessible for intratumoral injection. Tumor biopsies are not required in the expansion cohort.
4. Patients must be 18 years of age or older.
5. Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
6. Patients must meet the following laboratory criteria:

   1. Absolute neutrophil count ANC ≥1.5 x 109/L (≥1500/mm3)
   2. Platelet count ≥75 x 109/L (≥75,000/mm3)
   3. Hemoglobin ≥8.0 g/dL (≥4.96 mmol/L)
   4. Serum creatinine ≤1.5 x ULN or calculated 24-hour creatinine clearance ≥60 mL/minute
   5. Aspartate aminotransferase (AST) ≤2.5 x ULN; ALT ≤2.5 x ULN or AST/ALT <5 x ULN if liver involvement
   6. Total bilirubin ≤1.5 x ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin <3 mg/dL (51.3 μmol/L)
7. Women of childbearing potential and men must agree to use effective contraceptive methods from Screening throughout the study treatment period and until at least 4 weeks after the last dose of study drug.
8. Patients must be willing and able to provide signed informed consent and comply with the study protocol.

Exclusion Criteria:

1. Patients who have received prior therapy with a TLR agonist Patients who have received experimental vaccines or immune therapies other than PD-(L)1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors (e.g., Imlygic®) should be discussed with the Medical Monitor to confirm eligibility.

   Note: (prior treatment with a topical TLR agonist (e.g. imiquimod) is permitted).
2. Patients who have received treatment with IFN-α within the previous 6 months prior to enrollment.
3. Patients with known hypersensitivity to any oligodeoxynucleotide that cannot be adequately managed with appropriate prophylaxis; e.g. steroids.
4. Patients with active autoimmune disease requiring disease-modifying therapy.
5. Patients requiring concurrent systemic steroid therapy higher than physiologic dosage (>10mg/day of prednisone or equivalent).
6. Patients with another primary malignancy that has not been in remission for at least 3 years, unless approved by the Idera Medical Monitor. The following are exempt from the 3-year limit: non-melanoma skin cancer, curatively treated localized prostate cancer with non-detectable prostate-specific antigen, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou (Pap) smear, and thyroid cancer (except anaplastic).
7. Patients with active infections requiring systemic treatment.
8. Patients who are known to be hepatitis B surface antigen positive.
9. Patients with a known diagnosis of human immunodeficiency virus (HIV) infection.
10. Women who are pregnant or breastfeeding.
11. Patients with known central nervous system, meningeal, or epidural disease. Patients with stable brain metastases following definitive local treatment are eligible if steroid requirement is <10 mg/day of prednisone (or equivalent).
12. Patients with impaired cardiac function or clinically significant cardiac disease:

    1. New York Heart Association Class III or IV cardiac disease, including preexisting clinically significant ventricular arrhythmia, congestive heart failure, or cardiomyopathy
    2. Unstable angina pectoris ≤6 months prior to study participation
    3. Acute myocardial infarction ≤6 months prior to study participation
    4. Other clinically significant heart disease (i.e., Grade ≥3 hypertension, history of labile hypertension, or poor compliance with an anti-hypertensive regimen)
13. Have not recovered (to baseline or Grade ≤1) from toxicity associated with prior treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Dose Evaluation Cohorts, non-Melanoma Dose Evaluation Cohorts: Number of patients with treatment-related adverse events as assessed by CTCAE to determine the recommended Phase 2 dose (RP2D). | 51 weeks of treatment
Dose Evaluation Cohorts, non-Melanoma Dose Evaluation Cohorts: Objective response rate | Assessed every 6 weeks for duration of study participation, which is estimated to be 51 weeks
Melanoma Expansion Cohort: Objective response rate | Assessed every 9 weeks for duration of study participation, which is estimated to be 51 weeks
Melanoma Expansion Cohort: Number of patients with treatment-related adverse events as assessed by CTCAE | 51 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Idera Medical Director, Study Director — Idera Pharmaceuticals, Inc.
Locations (12):
- United States (8):
  - Scottsdale Healthcare Hospitals DBA Honor Health, Scottsdale, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Francisco (UCSF), San Francisco, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - St. Luke's Hospital, Easton, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - The Ella Lemelbaum Institute for Immuno-Oncology, Ramat Gan